CLINICAL TRIAL: NCT04352673
Title: Reliability of Elbow Flexion and Extension Strength Measurement Protocols Using a Hand-held Dynamometer
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Karabay, Research assistant, Dokuz Eylul University
Other Study IDs: 5001-GOA
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals: Healthy students 18 years and older
  Interventions: Diagnostic Test: Elbow flexion and extension strength measurements using a hand-held dynamometer

INTERVENTIONS:
Diagnostic Test: Elbow flexion and extension strength measurements using a hand-held dynamometer — Elbow flexion and extension strength of the participants will be measured in both arms in the supine, prone, and sitting positions using a hand-held dynamometer.

SUMMARY:
The aim of the study was to investigate the intra-rater and inter-rater reliability of elbow strength measurement procedures performed in different body postures and shoulder and elbow positions using a hand-held dynamometer in healthy individuals and to determine the standard error of measurement (SEM) and minimum detectable change (MDC) values for these procedures.

DETAILED DESCRIPTION:
Healthy university students aged 18 years and older will be included in the study. Elbow flexion and extension strength will be measured in both arms in different body postures and shoulder and elbow positions using a hand-held dynamometer. Thus, the reliability of these procedures will be investigated, and the standard error of the measurement and the minimum detectable change will be determined. Strength measurements will be performed by two physiotherapists on each arm of the participants and repeated between 3 - 7 days after the measurement to evaluate both intra-rater and inter-rater reliability.

3 different positions will be used for elbow flexion:

1. Participants sit on a stool, and their arms are at the side with the elbow flexed 90° (forearm in supination).
2. Participants sit on a stool, and their shoulder and elbow are flexed to 90° (forearm in supination) and supported on the treatment table.
3. Participants lie supine and place their shoulders on neutral position and elbow flexed 90° (forearm in supination).

3 different positions will be used for elbow extension:

1. Participants sit on a stool, and their shoulder and elbow are flexed to 90° (forearm in supination) and supported on the treatment table.
2. Participants lie supine and place their shoulders on neutral position and elbow flexed 90° (forearm in supination).
3. Participants lie prone, and their shoulders аre placed at 90° abduction and elbows flexed to 90°.

ELIGIBILITY:
Inclusion Criteria:

-Being older than 18 years old

Exclusion Criteria:

* Having neck, shoulder, elbow or forearm injuries in the last 6 months,
* Having upper extremity or neck fracture or surgical history
* Symptoms related to the neck, shoulder, elbow, and forearm at the time of assessment
* Having neurological or systemic musculoskeletal diseases or disorders
* Having a diagnosis of chest deformity or scoliosis
* Doing regular exercise related to upper extremity for the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students of Dokuz Eylul University, School of Physical Therapy and Rehabilitation
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Elbow flexion measurements | Measurements will be performed in two sessions (3-7 days between sessions)
  Elbow flexion strength will be measured in 3 different positions.
Elbow extension measurements | Measurements will be performed in two sessions (3-7 days between sessions)
  Elbow extension strength will be measured in 3 different positions.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi Yesilyaprak, PhD, Principal Investigator — Dokuz Eylul University; Fatma Özden, MS, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No